CLINICAL TRIAL: NCT03386123
Title: A Comparison of Cognitive Behaviour Therapy for Insomnia (CBTi) and Usual Audiological Rehabilitation in the Management of Tinnitus Related Insomnia
Brief Title: A Comparison of CBTi and Usual Treatment for Tinnitus Related Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: British Tinnitus Association (Other); University College, London (Other)
Responsible Party: Principal Investigator, Dr Laurence McKenna, Consultant Clinical Psychologist, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLondonH
Record Dates: First submitted 2017-12-08; First posted 2017-12-29 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Tinnitus; Insomnia
Keywords: Tinnitus; Insomnia; Cognitive Behaviour Therapy
MeSH Terms: conditions — Tinnitus; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behaviour Therapy for Insomnia (CBTi) (Experimental): A standard CBTi programme for the treatment of primary insomnia, with six, 2 hour, group sessions over eight weeks. There will be minor adaptations for tinnitus, including making specific reference to tinnitus and psycho-education about tinnitus. Every session concludes with provision of a homework task and a sleep diary to complete over the next week. The CBTi course will be supported by providing participants with a CD with some relaxation exercises and a booklet that covers the information given in the session.
  CBTi includes: Sleep restriction, stimulus control, Sleep hygiene, Relaxation training, Paradoxical intention, Cognitive therapy: Targeting unhelpful beliefs about sleep and worry, Behavioural experiments: Testing unhelpful beliefs and adjusting sleep related behaviour.
  Interventions: Behavioral: Cognitive Behaviour Therapy for Insomnia
- Standard Audiological Care (SAC) (Active Comparator): A group intervention that fits with reported audiological treatment of people with tinnitus and significant sleep impairment. This involves psycho-education about tinnitus, habituation, sleep and sleep hygiene. Relaxation will be advised and information provided. A bedside sound generator, as used in routine clinical practice will be provided. Information will be based on standard advice given by hearing therapists/audiologists and will not include specific psychological techniques which are not part of SAC. The group will be generally supportive.
  SAC tends not to involve repeated meetings; after the initial session, there will be one follow up session 8 weeks later. Follow up will allow for question and answer, and reports on what has been useful. Both sessions will last for 2 hours
  Interventions: Behavioral: Standard Audiological Care
- Sleep Support Group (SSG) (Placebo Comparator): Participants will meet in a group, which will offer equivalent contact with therapists and a supportive group milieu as CBTi. It will focus on the potential benefits of a supportive group and will not include specific advice.
  Participants will complete 2-week sleep diaries as baseline and outcome measures at the four time-points, which will be checked within the session to ensure that participants know how to complete them correctly. The SSG will meet in a group for six sessions, over eight weeks, each of 2 two hours duration.
  Interventions: Behavioral: Sleep Support Group

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy for Insomnia — Continuous maintenance of sleep diary, cognitive behaviour therapy, including cognitive restructuring, and behavioural change focusing on sleep restriction and safety behaviours.
  Arms: Cognitive Behaviour Therapy for Insomnia (CBTi)
Behavioral: Standard Audiological Care — Maintenance of sleep diary at key times. Psycho-education, provision of bedside sound generator.
  Arms: Standard Audiological Care (SAC)
Behavioral: Sleep Support Group — Maintenance of sleep diary at key times. Social support focused on tinnitus and sleep problems.
  Arms: Sleep Support Group (SSG)

SUMMARY:
There is evidence that CBT for insomnia (CBTi) is an effective treatment for sleep disturbance both as a primary problem and when co-morbid with other health problems, such as chronic pain.

This study will investigate the effectiveness of CBTi as a treatment for tinnitus related insomnia. Tinnitus patients reporting clinically significant insomnia will be offered sleep-specific treatment. Six sessions of CBTi will be offered to one group of patients and 2 sessions standard audiological care (psycho-education and sleep hygiene) will be offered to another group. Both groups will be offered sound enrichment at night. In order to take account of the possible effects of clinical contact a third group will be offered 6 sessions of support without a focused tinnitus or sleep intervention. Accepted measures of sleep disturbance will be used as well as measures of tinnitus complaint.

All treatment/contact will be provided at the Royal National Throat Nose & Ear Hospital. Participants will be involved in the study (inc. baseline period {2 weeks}, intervention {8 weeks} and follow-ups {4 and 20 weeks}) for 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least moderately distressing tinnitus (above a set minimum score on the Mini TQ) for at least six months and problematic insomnia (above a set minimum score on the Insomnia Severity Index (ISI) and for tinnitus related insomnia to be identified in clinical interview) as result of tinnitus, for at least three months.
* Patient wishes to work on improving sleep.
* Sufficient understanding of English and sufficient hearing ability to take part in for group discussions and to complete questionnaires.
* Patient has had tinnitus assessed by a doctor and an audiological specialist.
* Willing and able to provide written consent. Able to regularly attend clinic in London, United Kingdom.

Exclusion Criteria:

* • Organic sleep disorders present (e.g. Obstructive Sleep Apnoea, delayed phase sleep, etc.) assessed with a subscale of the hospital sleep unit's sleep disorder and snoring proforma.

  * Currently pregnant, planning pregnancy or breastfeeding.
  * Alcohol or drug dependent.
  * Currently suffering with severe mental illness (psychosis, severe anxiety or mood disorder).
  * Reports active risk to themselves or others. Still undergoing medical investigations into sleep and / or tinnitus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) score | At first and last treatment sessions and at 1 and 6 month follow-ups
  7-item questionnaire, each item rates 0 - 4. Total scores range from 0-28 with higher scores indicating more severity.
Change in the amount of sleep obtained | A 2-week sleep diary will be kept 2 weeks prior to the first and last treatment sessions and to the 1 and 6 month follow-ups.
  Average of all of the following metrics obtained from 2 weeks of sleep diary measure:
  Sleep Onset Latency - lower score indicates better sleep; Wake Time After Sleep Onset - lower score indicate better sleep; Number of night time awakenings - lower scores indicate better sleep; Total Sleep Time - higher scores indicate better sleep; Time in Bed - included only so that Sleep Efficiency can be calculated: Sleep Efficiency (Total Sleep Time / Time in Bed x 100) - higher scores indicate better sleep.
  Diary measures for sleep quality (0= worst possible to 10=best possible), tinnitus annoyance (0= not at all to 10= extremely), refreshed at waking (0= not at all to 10= very refreshed) and quality of day time functioning (0= very poor to 10= very good).

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index score | At first and last treatment sessions and at 1 and 6 month follow-ups
  10-item questionnaire. Sum of 7 components; global score range 0 - 21; higher scores indicate worse sleep quality.
Change in Dysfunctional Beliefs and Attitudes About Sleep Questionnaire - abbreviated version (DBAS-16) score | At first and last treatment sessions and at 1 and 6 month follow-ups
  16-item questionnaire scored on a 0-10 scale. The average score is calculated from all individual scores and ranges from 0-10; higher scores indicate more dysfunctional / unrealistic beliefs about / sleep.
Change in Tinnitus Catastrophizing Scale score | At first and last treatment sessions and at 1 and 6 month follow-ups
  13-item questionnaire scored on a 0-4 scale. Total sum of scores range from 0 - 52. Higher scores indicate higher levels of catastrophizing.
Mini Tinnitus Questionnaire score | Screening
  Construct: Tinnitus complaint 12-item questionnaire scored on a 0 - 2 scale. Total sum of scores range 0-24. Higher scores indicate presence of tinnitus. A score of 8 or more indicates the presence of a clinical level of tinnitus-related distress.
Change in the Tinnitus Questionnaire score | At first and last treatment sessions and at 1 and 6 month follow-ups
  Construct: Tinnitus complaint 41-item questionnaire scored on a 0 - 2 scale. Total sum of scores ranges from 0-82; higher scores indicate presence of tinnitus. The reliable change criterion is 11.08.
Change in subjective measure of tinnitus loudness | At first and last treatment sessions and at 1 and 6 month follow-ups
  Visual Analogue Scale from 0mm to 100mm; higher scores indicate greater loudness of tinnitus.
Change in Clinical Outcome in Routine Evaluation - Outcome Measure score | At first and last treatment sessions and at 1 and 6 month follow-ups
  Construct: general psychological distress 34-item questionnaire scored on a 0-4 scale. The average of all the scores is calculated and then multiplied by 10, so the scores can range from 0 to 40; a clinical cut-off score is 10 and clinically significant change is 5.
Change in Patient Health Questionnaire-9 score | At first and last treatment sessions and at 1 and 6 month follow-ups
  Construct: Depression 9-item questionnaire scored on a 0-3 scale; total sum of scores ranges from 0-27 with higher scores indicate greater depression severity.
Change in Generalized Anxiety Disorder Assessment-7 score | At first and last treatment sessions and at 1 and 6 month follow-ups
  7-items questionnaire scored on a 0-3 scale; total sum of scores ranges from total score range: 0-21 with higher score indicating more severe anxiety.
Change in EuroQOL score | At first and last treatment sessions and at 1 and 6 month follow-ups
  Construct: health status (dimensions: mobility, self-care, performing usual activities, pain or discomfort; anxiety or depression); each state is referred to in terms of a 5 digit code; The answers given to EQ-5D allow 243 unique health states to be identified and can be converted into EQ-5D index and utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analogue Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Change in Work and Social Adjustment Scale score | At first and last treatment sessions and at 1 and 6 month follow-ups
  Construct: impaired functioning 5-item questionnaire scored on a 0-8 scale; total sums of scores range from 0-40 with higher scores indicating greater functional impairment.
Satisfaction and feedback | At the end of treatment and at six month follow-up point
  Questionnaire asking individuals to rate the following on a 0 - 10 scale (from not at all to extremely) How useful was treatment? How relevant was treatment? How acceptable was treatment? They are also asked to provide qualitative feedback in the form of comments in response to questions about what changes they have noticed, what aspects of treatment were most and least useful, what they would have liked to be different and any other comments.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Laurence, PhD, Principal Investigator — UCLH
Locations (1):
- Uclh (Rntneh), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marks E, Hallsworth C, McKenna L. Cognitive behavioural therapy for insomnia (CBTi) as a treatment for tinnitus-related insomnia: protocol for a randomised controlled trial. Trials. 2019 Dec 2;20(1):667. doi: 10.1186/s13063-019-3778-5. PMID 31791396